CLINICAL TRIAL: NCT01956994
Title: The Effect of Whey Protein Supplementation on Cerebrovascular and Cognitive Function in Older Adults
Brief Title: The Effect of Whey Protein Supplementation on Vascular and Cognitive Function in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: Dairy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DRI-1154
Record Dates: First submitted 2013-08-26; First posted 2013-10-08 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Blood Pressure
Keywords: Whey Protein; Arterial Stiffness; Neurovascular Coupling; Cerebrovascular Reactivity; Hemodynamics; Blood Flow; Pulsatility
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whey protein supplement (Experimental): Subjects will be instructed to consume 40 g whey protein each day for 12 weeks.
  Interventions: Dietary Supplement: Whey protein supplement
- Carbohydrate supplement (Active Comparator): Subjects will be instructed to consume a carbohydrate supplement (iso-caloric to the whey supplement) each day for 12 weeks.
  Interventions: Dietary Supplement: Carbohydrate supplement

INTERVENTIONS:
Dietary Supplement: Whey protein supplement — Supplements will be provided in powder form and mixed into beverages to be consumed twice per day (after breakfast and after dinner).
  Other Names: 100% whey protein isolate
  Arms: Whey protein supplement
Dietary Supplement: Carbohydrate supplement — Supplements will be provided in powder form and mixed into beverages to be consumed twice per day (after breakfast and after dinner).
  Other Names: Maltodextrin
  Arms: Carbohydrate supplement

SUMMARY:
The "hardening of the arteries" observed with aging raises blood pressure and contributes to poor brain blood flow and loss of cognitive function (i.e. attention, memory, solving problems, making decisions). Cognition is the most important determinant of overall health status, quality of life, functional ability and independence in older adulthood. Nutraceutical strategies have received considerable attention as they may improve cardiovascular health with far fewer side effects compared to drugs. In this regard, dairy products are particularly attractive. Higher dairy consumption is associated with lower blood pressure and improved memory in adults. Milk proteins have natural blood pressure lowering effects. Studies conducted in animals have demonstrated that whey protein (a component of milk protein) may also increase artery elasticity. This is important given the strong association between artery elasticity, brain blood flow, and risk for cognitive decline.

The investigators propose to conduct a randomized double-blind placebo controlled study comparing the effects of whey protein supplementation or carbohydrate placebo on measures of artery elasticity, brain blood flow, and cognitive function in older adults. Whey protein may be a novel dietary therapy to improve both artery health and brain health in older adults.

DETAILED DESCRIPTION:
Participants will be randomly assigned to receive either 50 g whey protein isolate or placebo each day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ages of 60-85 years

Exclusion Criteria:

* acute or terminal illness
* Montreal Cognitive Assessment < 26 (indicating dementia)
* myocardial infarction or stroke in the previous 6 months or other symptomatic coronary or peripheral artery disease
* type I or type II diabetes mellitus
* visual impairment
* upper or lower extremity fracture in the previous 6 months
* uncontrolled hypertension (150/90 mm Hg)
* cigarette smoking
* chronic kidney disease (albumin/creatinine ratio (ACR) between 30-300 ug albumin/mg creatinine)
* liver disease
* chronic pulmonary/respiratory disease
* body mass index (kg/m2) < 21 or > 32
* recent weight loss or gain greater than 7.5% of body weight within the previous 6 months
* currently supplementing diet with whey protein products
* milk-protein allergy, or allergy to para-aminobenzoic acid (PABA)
* head injury or symptoms of concussion in the past 3 months

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in carotid artery blood pressure at 6 and 12 weeks | These outcomes will be assessed at baseline, 6-weeks and 12-weeks.

SECONDARY OUTCOMES:
Change in arterial stiffness at 6 and 12 weeks | These outcomes will be assessed at baseline, 6-weeks and 12-weeks.
Change in endothelial function at 6 and 12 weeks | These outcomes will be assessed at baseline, 6-weeks and 12-weeks.
Change in cognitive function at 6 and 12 weeks | These outcomes will be assessed at baseline, 6-weeks and 12-weeks.
Change in neurovascular coupling (carotid and cognitive perfusion during a mental challenge) at 6 and 12 weeks | These outcomes will be assessed at baseline, 6-weeks and 12-weeks.

OTHER OUTCOMES:
Change in physical activity at 6 and 12 weeks | These outcomes will be assessed at baseline, 6-weeks and 12-weeks.
Change in dietary patterns at 6 and 12 weeks | These outcomes will be assessed at baseline, 6-weeks and 12-weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin S Heffernan, Ph.D., Principal Investigator — Syracuse University
Locations (1):
- Syracuse University Human Performance Laboratory, Syracuse, New York, United States